CLINICAL TRIAL: NCT06015620
Title: CoMOrbidities Resolution After Mini-GAstric Bypass Surgery for Morbid Obesity and Change in BOdy Composition: A Prospective Cohort Study (MOGAMBO Study)
Brief Title: Comorbidities Resolution After MGB Surgery and Change in Body Composition
Acronym: MOGAMBO
Status: Recruiting | Type: Observational
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr. Prakash Kumar Sasmal, Additional Professor of General Surgery, All India Institute of Medical Sciences, Bhubaneswar
Other Study IDs: AIIMSBBSR/PGThesis/2023-24/61
Record Dates: First submitted 2023-08-22; First posted 2023-08-29 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Morbid Obesity; Type2diabetes; Sleep Apnea; Hypothyroidism; Hypertension; Lipid Disorder; Non-Alcoholic Fatty Liver Disease; Chronic Venous Hypertension With Ulcer
Keywords: morbid obesity; OSA; mini gastric bypass; metabolic surgery; polysomnography; metabolic syndrome; DEXA scan; bioelectrical impedance; body composition
MeSH Terms: conditions — Obesity, Morbid; Sleep Apnea Syndromes; Hypothyroidism; Hypertension; Lipid Metabolism Disorders; Non-alcoholic Fatty Liver Disease; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with morbid obesity undergoing metabolic surgery (Mini gastric bypass): The patients undergoing mini gastric bypass surgery for morbid obesity and its different comorbidities like type 2 diabetes, hypertension, dyslipidemia, obstructive sleep apnea, hypothyroidism and chronic venous hypertension.
  Interventions: Procedure: Mini gastric bypass surgery

INTERVENTIONS:
Procedure: Mini gastric bypass surgery — Mini gastric bypass surgery is a common metabolic or bariatric surgery done world wide for patients suffering from morbid obesity not managed by non surgical modalities of treatment.

SUMMARY:
This observational study aims to learn about the correlation between the improving comorbidities associated with obesity after MGB (Mini-Gastric Bypass) surgery and changes in body composition in morbidly obese patients. The main questions it aims to answer are:

To study the correlation between the improving comorbidities associated with obesity after MGB(Mini-Gastric Bypass) surgery and changes in body composition.

Other objectives are:

* Changes in the parameters of the metabolic syndrome after surgery
* Changes in the cardiovascular risk biomarkers after metabolic surgery
* Emergence in complications arising out of surgery requiring any intervention or causing a prolonged hospital stay, or requiring additional outpatient visits.

Type of Study: An observational study in which participants with morbid obesity will undergo mini-gastric bypass surgery as per routine protocol. No separate experimental interventions will be done in the study for the participants.

DETAILED DESCRIPTION:
Evidence supports that bariatric or metabolic surgery is more effective than conventional therapy in controlling obesity and its related comorbidities. Although bariatric surgery has been widely practised for many years worldwide, there is still a need to understand the correlation between improving comorbidities associated with morbid obesity and body composition change post-surgery. Amongst the comorbidities, type II diabetes, sleep apnea, hypertension, and hypothyroidism are the significant ones associated with morbid obesity. A disturbed quality of sleep results in daytime sleepiness, cardiac problems, renal problems, etc., which in turn grossly reduces the work efficiency of an individual and increases morbidity and mortality. From our experience, after a metabolic surgery (mini-gastric bypass -MGB), the investigators find comorbidities, especially sleep apnoea and type II diabetes, getting controlled early before significant weight loss has started. Also, there is an improvement in the parameters of the metabolic syndrome after metabolic surgery. The prospective cohort study aims to correlate the comorbidities resolution after mini-gastric bypass surgery for morbid obesity and change in body composition.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing laparoscopic MGB surgery for morbid obesity and it's associated comorbidities

Exclusion Criteria:

* Patients not giving consent for the study
* All patients who were undergoing a redo-procedure for recurrence were excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from morbid obesity and its associated comorbidities like type 2 diabetes, hypertension, obstructive sleep apnea, hypothyroidism, dyslipidemia and chronic venous hypertension of the legs with its complications.
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
To study the correlation between the improving comorbidities associated with obesity after MGB(Mini-Gastric Bypass) surgery and changes in body composition. | 3 years
  The comorbidities associated with obesity like type2 diabetes, sleep apnea, dyslipidemia, hypothyroidism and other components of metabolic syndrome improves way ahead after the metabolic surgery as compared to an expected change in the body composition. This study will bring out the correlation between the change in body composition and the morbidity resolution.

SECONDARY OUTCOMES:
Changes in the parameters of the metabolic syndrome after surgery | 3 years
  Components of the metabolic syndrome improve after metabolic surgery after different timelines. This study will bring out the time line of resolution of comorbidities after a metabolic surgery.
Changes in the cardiovascular risk biomarkers after metabolic surgery | 3 years
  Cardiovascular biomarkers like C reactive proteins (CRP) is stated to improve over time after a metabolic surgery. This study will find out the improvement in the CVS biomarker after the metabolic surgery.
Emergence in complications arising out of surgery requiring any intervention or causing a prolonged hospital stay, or requiring additional outpatient visits | 3 years
  The mini gastric bypass surgery done for morbid obesity is a malabsorption procedure done in patients suffering from morbid obesity. Expected changes in the post-operative patients are protein-energy malnutrition, essential vitamins like B12, D, etc, and mineral deficiency may occur. So a follow up of the patients in the post operative period will reveal any postoperative nutritional changes and there consequences.

CONTACTS AND LOCATIONS:
Overall Officials: Prakash K Sasmal, MS, FACS, Principal Investigator — All India Institute of Medical Sciences, Bhubaneswar, India
Locations (1):
- All India Institute of Medical Sciences, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No
Only the result of the study will be provided at the end. No individual patients detail will be revealed. However, the statistical analysis details, including the study protocol can be shared if required by any researcher.

REFERENCES:
- [Background] Rudnicki Y, Slavin M, Keidar A, Kent I, Berkovich L, Tiomkin V, Inbar R, Avital S. The effect of bariatric surgery on hypothyroidism: Sleeve gastrectomy versus gastric bypass. Surg Obes Relat Dis. 2018 Sep;14(9):1297-1303. doi: 10.1016/j.soard.2018.06.008. Epub 2018 Jun 15. PMID 30049595
- [Result] Achamrah N, Colange G, Delay J, Rimbert A, Folope V, Petit A, Grigioni S, Dechelotte P, Coeffier M. Comparison of body composition assessment by DXA and BIA according to the body mass index: A retrospective study on 3655 measures. PLoS One. 2018 Jul 12;13(7):e0200465. doi: 10.1371/journal.pone.0200465. eCollection 2018. PMID 30001381
- [Result] Ravesloot MJ, Hilgevoord AA, van Wagensveld BA, de Vries N. Assessment of the effect of bariatric surgery on obstructive sleep apnea at two postoperative intervals. Obes Surg. 2014 Jan;24(1):22-31. doi: 10.1007/s11695-013-1023-y. PMID 23856989
- [Result] Fritscher LG, Canani S, Mottin CC, Fritscher CC, Berleze D, Chapman K, Chatkin JM. Bariatric surgery in the treatment of obstructive sleep apnea in morbidly obese patients. Respiration. 2007;74(6):647-52. doi: 10.1159/000107736. Epub 2007 Aug 29. PMID 17728530
- [Result] Cogollo VJ, Rivera CE, Valera RJ, Sarmiento-Cobos M, Montorfano L, Wasser E, Lo Menzo E, Szomstein S, Rosenthal RJ. Improvement of glucose metabolism following rapid weight loss after bariatric surgery and its impact on reduction of visceral abdominal fat versus free fat muscle. Surg Obes Relat Dis. 2021 May;17(5):933-938. doi: 10.1016/j.soard.2021.01.031. Epub 2021 Feb 2. PMID 33715992
- [Result] Snelder SM, Pouw N, Aga Y, Castro Cabezas M, Biter LU, Zijlstra F, Kardys I, van Dalen BM. Cardiovascular Biomarker Profiles in Obesity and Relation to Normalization of Subclinical Cardiac Dysfunction after Bariatric Surgery. Cells. 2022 Jan 26;11(3):422. doi: 10.3390/cells11030422. PMID 35159232
- [Result] Castanha CR, Tcbc-Pe AABF, Castanha AR, Belo GQMB, Lacerda RMR, Vilar L. Evaluation of quality of life, weight loss and comorbidities of patients undergoing bariatric surgery. Rev Col Bras Cir. 2018 Jul 16;45(3):e1864. doi: 10.1590/0100-6991e-20181864. English, Portuguese. PMID 30020323